CLINICAL TRIAL: NCT04550741
Title: Long-term Maintenance Benefits of a Pulmonary Rehabilitation Program Using a Mobile Digital Solution: a Prospective, Randomized, Controlled, Multicenter Study in a Population of COPD Patients
Acronym: m-Rehab COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL17_0030; 2017-A01248-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-06-29; First posted 2020-09-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Telerehabilitation; Telemedicine; Exercise training; Quality of life; E-health; Connected objects; Care manager
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Telerehabilitation

STUDY DESIGN:
Masking Description: This study will be an Open study.
  For the primary outcome the analysis will be blind to the investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation (Experimental): Experimental group of 100 patients using the M-Réhab BPCO telerehabilitation solution. The solution will be provided during the fourth and final week of RR's stay during which patients will be trained to use all of the solution's features. Patients will carry out the entire post-rehabilitation using the remote rehabilitation solution and will benefit from medical assessments by teleconsultation at 1, 3, 6 and 12 months as well as assessments at 3, 6 and 12 months by filling. electronic auto-questionnaires followed by a telephone quality control if necessary. A final evaluation at 12 months, by videoconference, will be carried out at the patient's home.
  Interventions: Other: telerehabilitation
- Standard chronic care (No Intervention): following usual standard chronic care. Patients will receive during the last week of stay in the center, the usual advice to continue physical activity and nutritional advice at home. The evaluations at 3, 6 and 12 months will be done by electronic filling of auto-questionnaires followed by a telephone quality control if necessary. A final evaluation at 12 months, by videoconference, will be carried out at the patient's home.

INTERVENTIONS:
Other: telerehabilitation — After obtaining consent, the volunteers will be included in the study at the start of the 4th week and randomized into two arms: Experimental and Control group
  Other Names: Digital solution of telerehabilitation with remote connected objects
  Arms: Telerehabilitation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a public health problem: high prevalence; increasing morbidity and mortality; impact on health costs. Pulmonary rehabilitation (PR) is a multidisciplinary intervention combining exercise training, therapeutic education, psychosocial and behavioral interventions. Its effects are beneficial in the short and medium terms but are limited in time, between 6 and 12 months, for patients who do not pursue regular physical activity (PA) in post-rehabilitation and who do not adopt behavioral changes for health, by loss of motivation. Maintaining the long-term benefits acquired during a short-term PR program is therefore a major issue in the management of COPD. The recent development of remote rehabilitation is a promising approach that has been studied in few studies.

In a randomized, controlled and multicenter study, we propose to test the hypothesis that the use of a mobile telerehabilitation solution will allow COPD patients to mainain at long-term the benefits acquired during a short-temr programm and therfore improve their quality of life.

(PA) in post-rehabilitation and who do not adopt behavioral changes for health, by loss of motivation. Maintaining the long-term benefits acquired during a short-term PR program is therefore a major issue in the management of COPD. The recent development of remote rehabilitation is a promising approach that has been studied in few studies.

In a randomized, controlled and multicenter study, we propose to test the hypothesis that the use of a mobile telerehabilitation solution will allow COPD patients to mainain at long-term the benefits acquired during a short-temr programm and therfore improve their quality of life.

DETAILED DESCRIPTION:
Exclusion criteria:

* Presence of contraindications for exercise training (neuromuscular disease, orthopedic cause).
* Patients with significant and unstable cardiovascular disease.
* Inability to understand and/or answer questionnaires.
* Refusal to use a smartphone or digital device.
* Unable to access an internet connection at home.

Analysis:

* The main analysis will be the univariate intention-to-treat analysis of the primary outcome.
* Secondary analyzes will include:
* Analysis with intention to treat secondary endpoints.
* Multivariate analysis of the efficiency criteria.
* Univariate and multivariate medico - economic cost - utility analyzes, with their respective sensitivity analyzes.

Protocol:

This prospective, randomized study with two parallel arms, controlled against standard chronic care will be multicentric and open.

* Patients included will be patients diagnosed with COPD who are on RR for four weeks in one of the three centers participating in the study.
* Participation in the study will be offered after verification of the eligibility criteria, during the 3rd week of the stay.
* The information note will then be provided to them.
* After obtaining consent, the volunteers will be included in the study at the start of the 4th week and randomized into two arms:
* - Experimental group of 100 patients using the M-Réhab BPCO telerehabilitation solution. The solution will be provided during the fourth and final week of RR's stay during which patients will be trained to use all of the solution's features. Patients will carry out the entire post-rehabilitation using the remote rehabilitation solution and will benefit from medical assessments by teleconsultation at 1, 3, 6 and 12 months as well as assessments at 3, 6 and 12 months by filling. electronic auto-questionnaires followed by a telephone quality control if necessary. A final evaluation at 12 months, by videoconference, will be carried out at the patient's home.
* Control group of 100 patients following usual standard chronic care. Patients will receive during the last week of stay in the center, the usual advice to continue physical activity and nutritional advice at home. The evaluations at 3, 6 and 12 months will be done by electronic filling of auto-questionnaires followed by a telephone quality control if necessary. A final evaluation at 12 months, by videoconference, will be carried out at the patient's home.

The duration of the inclusions is 18 months and the follow-up will be carried out over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD according to the GOLD (Global Initiative for Chronic Obstructive Lung Disease) creteria.
* Presence of an incompletely reversible obstructive ventilatory disorder defined by a report VEMS / CVF lower than the lower limit of normal post-bronchodilator.
* Patient on RR for four weeks in respiratory rehabilitation center.
* Aged between 40 and 78 years.

Exclusion Criteria:

* Presence of contraindications for exercise training (neuromuscular disease, orthopedic cause).
* Patients with significant and unstable cardiovascular disease.
* Inability to understand and/or answer questionnaires.
* Refusal to use a smartphone or digital device.
* Unable to access an internet connection at home.

Ages: 40 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Quality of Life of chronic obstructive pulmonary disease patients after a 1-year téléherabilitaion versus standard care program, after an initial short-term pulmonary rehabilitation program | 12 months
  Quality of life assessed by the Saint Georges Respiratory Questionnaire. Three scores are calculated for the components: Symptoms; Activities; Impacts. A Total SCORE is also calculated.
  The minimum significant difference is 4 points.

SECONDARY OUTCOMES:
Pre-intentional variables | baseline
  Perceived risk: questionnaire focused on respiratory disease and conditioned by absence of adoption of physical activity behavior.
  Expectation of conséquences: questionnaire of the expected effects of Physical activity on physical health and psychological well-being.
  Self-efficacy: questionnaire relating to their perceived ability to perform the quantity of physical activity recommended by healthcare professionals.
  Intentions: determination and realization of physical activity behavior in the next months.
Post-intentional variables | 6 months
  planning: by a Questionnaire relating to the anticipation of the conditions to realize physical activity.
  self-efficacy with regard to barriers: questionnaire relating to their perceived ability to perform physical activity recommended despite the difficulties encountered.
  Social support:questionnaire relating to the behavior of the entourage habits: questionnaire on automatic nature of physical activity behavior.
Physical Activity behaviors. | 12 months
  Measured by the International Physical Activity Questionnaire as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
  walking consider to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS.
Predictive model of physical activity behavior | At 12 months
  Test a predictive model of physical activity behavior at 12 months in each of the two arm groups.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre hopsitalier universitaire de Montpellier, Montpellier, Occitanie
  - Clinique du Souffle, Osséja

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633